CLINICAL TRIAL: NCT02396030
Title: Effectiveness and Safety of 1g/Hour vs. 2g/Hour of Magnesium Sulfate Maintenance Dose for Eclampsia Prevention: Randomized Clinical Trial
Brief Title: Different Schemes of Magnesium Sulfate for Preeclampsia
Acronym: MGSO4
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After recommendation because of the impossibility to end study with 1 center only. Outcomes of patients already included will be evaluated.
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, MD PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MGSO4-2015
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate; nickelboussingaultite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulfate 50% - 1g/h (Active Comparator): After loading dose of 6g of magnesium sulfate, patients will receive the maintenance dose of 1g/hour of intravenous magnesium sulfate, for 24 hours
  Interventions: Drug: Magnesium sulfate 50% - 1g/h
- Magnesium sulfate 50% - 2g/h (Experimental): After loading dose of 6g of magnesium sulfate, patients will receive the maintenance dose of 2g/hour of intravenous magnesium sulfate, for 24 hours
  Interventions: Drug: Magnesium sulfate 50% - 2g/h

INTERVENTIONS:
Drug: Magnesium sulfate 50% - 1g/h — Patients will receive after the loading dose os magnesium sulfate, the maintenance dose of 1g/hour of intravenous of magnesium sulfate for 24 hours after loading dose
  Other Names: Mg SO4
  Arms: Magnesium sulfate 50% - 1g/h
Drug: Magnesium sulfate 50% - 2g/h — Patients will receive after the loading dose os magnesium sulfate, the maintenance dose of 1g/hour of intravenous of magnesium sulfate for 24 hours after loading dose
  Other Names: MgSO4
  Arms: Magnesium sulfate 50% - 2g/h

SUMMARY:
Eclampsia is an obstetric emergency capable of prophylaxis. To prevent and control seizures, there is no doubt that the magnesium sulfate (MgSO4) is the ideal drug. However, there are still questions regarding its use and dose. The scheme and the optimal time of administration remain to be elucidated. The objective of this trial is to compare the effectiveness and safety of intravenous magnesium sulfate in the maintenance phase 1g / h versus 2 g / h to prevent eclampsia in pregnant and postpartum women with severe preeclampsia (pure or superimposed).

DETAILED DESCRIPTION:
Hypertensive disorders are frequent during the course of pregnancy-puerperal cycle and an important cause of maternal morbidity and mortality, fetal and perinatal. The high frequency of maternal death can be explained by the presence of numerous complications such as eclampsia. Eclampsia is an obstetric emergency capable of prophylaxis. To prevent and control seizures, there is no doubt that the magnesium sulfate (MgSO4) is the ideal drug. However, there are still questions regarding its use and dose. The scheme and the optimal time of administration remain to be elucidated. Currently, allows the use of either 1 g / h to 2 g / h of magnesium sulphate during the maintenance phase to prevent eclamptic convulsions. However, there is no report in the literature of randomized controlled trials comparing different doses of magnesium sulfate in the maintenance phase to prevent eclampsia.

The objective of this study is to compare the effectiveness and safety of intravenous magnesium sulfate in the maintenance phase 1g / h versus 2 g / h to prevent eclampsia in pregnant and postpartum women with severe preeclampsia (pure or superimposed).There will be a trial randomized and triple blind in the Integrative Medicine Institute Prof. Fernando Figueira (IMIP) from March 2015 to April 2017, and will be included 2000 women randomized into two groups: MgSO4 maintenance dose of 1 g / h or 2 g / h. Patients who had eclampsia before loading dose, with use of other medications or illicit drugs that may interfere with maternal hemodynamics or with contraindications to the use of magnesium sulfate will be excluded. The primary endpoint will be the incidence of eclampsia. Other complications such as oliguria, bleeding, recurrence of seizures, disseminated intravascular coagulation, maternal death, presence of side effects related to the use of MgSO, neonatal outcome and other variables will be considered secondary outcomes. Randomization for preventive treatment of eclamptic seizures with MgSO4 1g / h or MgSO4 2g / h will be held according to a table of sequential numbers from one to 2000, using the letters A and B and not knowing its meaning. The analysis will be performed with the groups identified as A or B, breaking the secrecy only after the results obtained and prepared the tables, or by resolution of the External Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Severe Preeclampsia (pure and superimposed)

Exclusion Criteria:

* Eclampsia before administration of the loading dose of MgSO4 ;
* Use of other medications or illicit drugs that may interfere with maternal hemodynamics;
* Contraindications to the use of magnesium sulfate: known hypersensitivity to the drug, oliguria with urine output below 25 ml per hour or anuria (urine output absent) and myasthenia gravis.
* Use of mechanical ventilation

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ECLAMPSIA | From end of loading dose, until 24 hours after delivery
  Seizures that occur after the loading dose, during magnesium sulfate, until 24 hours after the delivery of the baby

SECONDARY OUTCOMES:
Placental abruption | From end of loading dose, until delivery of the child
  Occurence of placental abruption
postpartum hemorrhage | From end of loading dose, until 48 hours after delivery
  Occurence of postpartum hemorrhage, diagnosed clinically by the attending phisician
COMPLICATIONS | From end of loading dose, until 3 hours after delivery
  Occurence of a retained placenta
thromboembolic complications | From end of loading dose, until 15 days after delivery
  Diagnosis of thromboembolic complications bay doppler compression ultrasound or CT
liver failure | From end of loading dose, until 15 days after delivery
  Occurence of liver failure according to laboratorial exams
OLIGURIA | From end of loading dose, until 15 days after delivery
  Oliguria diagnosed as the presence of urine output under 0.5 (mililiters per kilogram) mL/kg for six hours,
RENAL FAILURE | From end of loading dose, until 15 days after delivery
  Occurence of renal failure diagnosed as the presence of oliguria for more than 24 hours or elevation serum creatinine (3X )
Disseminated intravascular coagulation (DIC) | From end of loading dose, until 15 days after delivery
  Presence of disseminated intravascular coagulation
acute pulmonary edema | From end of loading dose, until 15 days after delivery
  Presence of clinically diagnosis of acute pulmonary edema
Maternal death | From end of loading dose, until 42 days after delivery
  Maternal death occuring for direct obstetric causes
Composite maternal morbidity | From end of loading dose, until 42 days after delivery
  Presence of one of the investigated complications
RECURRENCE | From end of loading dose, until 24 hours after delivery
  Recurrence of seizures after loading dose of magnesium sulfate
additional anticonvulsant | From end of loading dose, until 24 hours after delivery
  Need for additional anticonvulsant after the use of magnesium sulfate
SIDE EFFECTS | From end of loading dose, until 24 hours after delivery
  Presence of side effects of magnesium sulfate use
DISCONTINUATION OF MAGNESIUM SULFATE | From end of loading dose, until 24 hours after delivery
  Occurence of discontinuation of treatment due to side effects
GLUCONATE USE | From end of loading dose, until 24 hours after delivery
  Need for the use of calcium gluconate
MAGNESIUM LEVELS | From end of loading dose, until 24 hours after delivery
  Serum magnesium levels evaluated at the beginning of maintenance dose and after 30. minutes, every 2 hours for six hours and after every six hours until 24 hous after loading dose.
  This outcome will be evaluated in the first 62 patients
Hypertensive crises | From end of loading dose, until 24 hours after delivery
  Presence of hypertensive crises and need for antihypertensive drugs and need to continue therapy for more than 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037